CLINICAL TRIAL: NCT05130879
Title: Evaluation of Building Resilience at Work (BRAW) Training Among Healthcare Workers: A Sequential Mixed Methods Design
Brief Title: Building Resilience @ Work Training Among Healthcare Workers
Acronym: BRAW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Lau Ying, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WF19-14
Record Dates: First submitted 2021-11-10; First posted 2021-11-23 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Resilience, Psychological
Keywords: Resilience training, Healthcare Workers

STUDY DESIGN:
Intervention Model Description: 1:1
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Research assistants and participants will be blinded to the conditions until baseline assessments (referring to the set of questionnaires they have to complete before starting the training) are completed, at which time a random number sequence in a excel file will be opened to reveal whether they will be in the intervention or waitlist condition. Participants will not be explicitly told of participants' study condition; however, they need to participate in the intervention, so full blinding is not possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRAW intervention group (Experimental): BRAW is designed as an online intervention comprising of six sessions over six weeks. The six sessions are: (1) happiness and positivity, (2) cognitive restructuring, (3) behavioural activation, (4) emotion regulation, (5) positive work climate and (6) problem solving.
  Interventions: Behavioral: BRAW
- Waitlist control group (No Intervention): Participants will receive the intervention after the follow-up assessment.

INTERVENTIONS:
Behavioral: BRAW — Sessions
  1. Happiness and positivity Understanding strengths and resilience and positive attitude
  2. Cognitive restructuring Identification dysfunctional automatic thoughts in problematic and emotional arousing situations Usage of cognitive -behavioural techniques to evaluate and modify dysfunctional thoughts and beliefs
  3. Behavioural activation Initiation and utilization of behavioural activation techniques for positive change by increasing pleasant events Healthy interpersonal relationships Importance of peer support
  4. Emotion regulation Preventing and managing conflict Emotion regulation abilities
  5. Positive work climate Building supportive work environment Development of supportive collegial relationships Promotion of coworker support
  6. Problem solving Problem-solving work-life problems Work-life balance Bringing it together
  Arms: BRAW intervention group

SUMMARY:
Background Given that the challenges in adjusting to shifting work, physical workload and high-strung nature, healthcare workers often encounter high stress, emotional exhaustion, low empathy, fatigue and burnout, which, in turn, result in sickness, absence, and high turnover. Hence, building resilience for future adversity among healthcare workers in the workplace is necessary.

Objectives To evaluate the effectiveness of the Building Resilience at Work (BRAW) on resilience, job engagement, intention to leave, employability, and work performance To explore healthcare workers' experience of the BRAW intervention.

Methods This study will evaluate the effectiveness of BRAW using a sequential mixed methods design in two phases. In phase I, a two-armed randomized controlled trial will be conducted to compare resilience, work engagement, coping skills, job satisfaction and life satisfaction with a waiting list control condition among 410 healthcare workers.

In phase II, the investigators will conduct a virtual individual interview to explore experiences on usability and acceptability after receiving the BRAW intervention using a sample of 33 healthcare workers.

Significance of research Considering the multifactorial and complexity of resilience at work in an increasingly dynamic healthcare environment, the content of resilience training can promote resilience, work engagement, coping skills, job satisfaction and life satisfaction among healthcare workers in order to reduce the turnover rate among healthcare workers in Singapore.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers aged 21 years or older
* Can read English
* Own and regularly use smartphone, tablet, laptop or desktop
* Can access the internet

Exclusion Criteria:

* Previous diagnosis of psychosis, severe depression, personality disorder and substance abuse at any point in their life

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
Resilience | Baseline
  A 6-item Brief Resilience Scale (BRS) is used to assess the ability to recover from stress. Items are rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). The total score ranges from 6 to 30, with higher scores signifying greater bounce-back resilience. BRS has demonstrated good reliability and validity.
Resilience | at 6 weeks
  A 6-item Brief Resilience Scale (BRS) is used to assess the ability to recover from stress. Items are rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). The total score ranges from 6 to 30, with higher scores signifying greater bounce-back resilience. BRS has demonstrated good reliability and validity.
Resilience | 12 weeks after training completes
  A 6-item Brief Resilience Scale (BRS) is used to assess the ability to recover from stress. Items are rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). The total score ranges from 6 to 30, with higher scores signifying greater bounce-back resilience. BRS has demonstrated good reliability and validity.

SECONDARY OUTCOMES:
Work engagement | Baseline
  A 9-item Utrecht Working Engagement Scale short version (UWES-9) is used to measure the participant's feelings in the context of work. Participant rate how often they experience these feelings on a 4-point Likert scale from 1 (never) to 4 (always). The total score ranges from 9 to 36 and higher scoring on UWES-9 indicates more work engagement. UWES-9 has confirmed satisfactory validity and reliability.
Work engagement | at 6 weeks
  A 9-item Utrecht Working Engagement Scale short version (UWES-9) is used to measure the participant's feelings in the context of work. Participant rate how often they experience these feelings on a 4-point Likert scale from 1 (never) to 4 (always). The total score ranges from 9 to 36 and higher scoring on UWES-9 indicates more work engagement. UWES-9 has confirmed satisfactory validity and reliability.
Work engagement | 12 weeks after training completes
  A 9-item Utrecht Working Engagement Scale short version (UWES-9) is used to measure the participant's feelings in the context of work. Participant rate how often they experience these feelings on a 4-point Likert scale from 1 (never) to 4 (always). The total score ranges from 9 to 36 and higher scoring on UWES-9 indicates more work engagement. UWES-9 has confirmed satisfactory validity and reliability.
Intention to leave | Baseline
  12-item Anticipated Turnover Scale (ATS)49 is used to measure intention to leave. Questions are related to one's anticipated length of time before leaving and certainty of leaving the job. Items are rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). The total score ranges from 12 to 60, with higher scores reflecting higher degree of turnover. CVI was 0.80-0.95 for items. Cronbach's alphas were 0.85-0.94 in several researches. Test-retest reliability coefficient was 0.84 in 2 weeks' interval.
Intention to leave | at 6 weeks
  12-item Anticipated Turnover Scale (ATS)49 is used to measure intention to leave. Questions are related to one's anticipated length of time before leaving and certainty of leaving the job. Items are rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). The total score ranges from 12 to 60, with higher scores reflecting higher degree of turnover. CVI was 0.80-0.95 for items. Cronbach's alphas were 0.85-0.94 in several researches. Test-retest reliability coefficient was 0.84 in 2 weeks' interval.
Intention to leave | 12 weeks after training completes
  12-item Anticipated Turnover Scale (ATS)49 is used to measure intention to leave. Questions are related to one's anticipated length of time before leaving and certainty of leaving the job. Items are rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). The total score ranges from 12 to 60, with higher scores reflecting higher degree of turnover. CVI was 0.80-0.95 for items. Cronbach's alphas were 0.85-0.94 in several researches. Test-retest reliability coefficient was 0.84 in 2 weeks' interval.
Employability | Baseline
  A 11-item Self-perceived Employability Scale (SPE) is used to assess employability. Participants are required to state their agreement with the items by selecting a number on a 5-point scale, from 1 (strong disagreement) to 5 (strong agreement). The total score ranges from 11 to 55, with higher score indicating perceived better employability. SPE has reported good internal consistency
Employability | at 6 weeks
  A 11-item Self-perceived Employability Scale (SPE) is used to assess employability. Participants are required to state their agreement with the items by selecting a number on a 5-point scale, from 1 (strong disagreement) to 5 (strong agreement). The total score ranges from 11 to 55, with higher score indicating perceived better employability. SPE has reported good internal consistency
Employability | 12 weeks after training completes
  A 11-item Self-perceived Employability Scale (SPE) is used to assess employability. Participants are required to state their agreement with the items by selecting a number on a 5-point scale, from 1 (strong disagreement) to 5 (strong agreement). The total score ranges from 11 to 55, with higher score indicating perceived better employability. SPE has reported good internal consistency
Work performance | Baseline
  A 18-item Individual Work Performance Questionnaire (IWPQ) is used to measure individual work performance. The IWPQ has a recall period of 3 months and a rating scale from 0 (seldom/never) to 4 (always/often) for task, contextual performance and counterproductive work behaviour. A mean score is calculated by adding the item scores, and dividing their sum by the number of items that range between 0 and 4, with higher scores reflecting higher individual work performance. The psychometric properties of the IWPQ indicated excellent internal consistency and good validity.
Work performance | at 6 weeks
  A 18-item Individual Work Performance Questionnaire (IWPQ) is used to measure individual work performance. The IWPQ has a recall period of 3 months and a rating scale from 0 (seldom/never) to 4 (always/often) for task, contextual performance and counterproductive work behaviour. A mean score is calculated by adding the item scores, and dividing their sum by the number of items that range between 0 and 4, with higher scores reflecting higher individual work performance. The psychometric properties of the IWPQ indicated excellent internal consistency and good validity.
Work performance | 12 weeks after training completes
  A 18-item Individual Work Performance Questionnaire (IWPQ) is used to measure individual work performance. The IWPQ has a recall period of 3 months and a rating scale from 0 (seldom/never) to 4 (always/often) for task, contextual performance and counterproductive work behaviour. A mean score is calculated by adding the item scores, and dividing their sum by the number of items that range between 0 and 4, with higher scores reflecting higher individual work performance. The psychometric properties of the IWPQ indicated excellent internal consistency and good validity.
Usage and satisfaction of training | at 6 weeks
  Usage is defined as an encompassing engagement, i.e., the time (in minutes) spent browsing the website and practicing the assigned homework in the previous weeks. Computer-generated indicators include the following: (1) session completion, (2) number of website visits, and (3) time spent on the website. At the end of the six-week program, attitude toward and satisfaction with the online training will be assessed using the self-developed eight-item usage and satisfaction of training. Each item is rated on a 4-point Likert scale from 1 to 4, and response options differed for the various items. The total score ranges from 8 to 32, and a high score represents better satisfaction of training. In addition, we have four open questions to obtain suggestions for improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Lau, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Ying Lau, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lau Y, Choi KC, Wong SH, Ang WW, Ang WHD, Lau ST. A randomized controlled trial investigating digital resilience training for healthcare professionals. Sci Rep. 2025 Dec 24;15(1):44514. doi: 10.1038/s41598-025-28028-z. PMID 41444278
- [Derived] Ang WHD, Lim ZQG, Lau ST, Dong J, Lau Y. Unpacking the Experiences of Health Care Professionals About the Web-Based Building Resilience At Work Program During the COVID-19 Pandemic: Framework Analysis. JMIR Med Educ. 2024 Jan 31;10:e49551. doi: 10.2196/49551. PMID 38294866